CLINICAL TRIAL: NCT02800642
Title: A Multi-center, Single-arm, Interventional Phase 4 Study to Evaluate a Treat and Extend Regimen of Intravitreal Aflibercept for Treatment of Macular Edema Secondary to Central Retinal Vein Occlusion
Brief Title: Evaluation of a Treat and Extend Regimen of Intravitreal Aflibercept for Macular Edema Secondary to CRVO
Acronym: CENTERA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17514; 2014-003193-17 (EudraCT Number)
Record Dates: First submitted 2016-06-10; First posted 2016-06-15 (Estimated); Results first posted 2020-07-08 (Actual); Last update posted 2020-07-08 (Actual); Status verified 2020-06

CONDITIONS: Central Retinal Vein Occlusion
Keywords: Bayer; Aflibercept; Eylea; Intravitreal
MeSH Terms: conditions — Retinal Vein Occlusion | interventions — aflibercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Intravitreal (IVT) aflibercept (Experimental): Participants with macular edema secondary to CRVO were treated with the study drug intravitreal aflibercept
  Interventions: Drug: Aflibercept (Eylea, BAY86-5321)

INTERVENTIONS:
Drug: Aflibercept (Eylea, BAY86-5321) — The recommended dose for intravitreal aflibercept was 2 mg equivalent to 50 μL. Study treatment was administered at baseline and at monthly intervals until stabilization of disease. When stability was achieved, the treatment interval could be extended based on visual and anatomic outcomes as judged by the treating investigator.

SUMMARY:
Central retinal vein occlusion (CRVO) occurs when the main blood vessel that transports blood away from the retina (the very back portion of the eye) becomes blocked, causing the leakage of fluid into the retina and thereby causing a swelling of the macula (the portion of the retina responsible for fine vision). This swelling is called macular edema. When the macula swells with fluid, central vision becomes blurry. The study drug aflibercept has been shown to reduce the amount of fluid and blood leaked into the retina. It can help to stabilize, and in many cases, improve the vision loss related to CRVO. Aflibercept has been approved for the treatment of macular edema secondary to CRVO in the United States (US), European Union (EU), Japan, and other countries.

The study was considered research because, although the study drug was already on the market for macular edema secondary to CRVO, there were no studies available that addressed the questions of what were useful intervals for treating and assessing patients, how did they differ among patients, and how were criteria applied for retreatment. The purpose of this study was to evaluate the effectiveness, treatment interval, and safety of the treatment regimen (pattern for administering treatment) in subjects with macular edema secondary to CRVO. In addition, this study explored new imaging methods for assessing the affected eye.

ELIGIBILITY:
Inclusion Criteria:

* Center-involved macular edema secondary to CRVO for no longer than 3 months (at the screening visit it should be ensured that the subjects will comply with the criterion of ≤ 3 months since onset of macular edema at their scheduled baseline visit).
* Adult subjects diagnosed with macular edema secondary to CRVO who are scheduled to be treated with IVT aflibercept as per investigator's routine treatment practice with the intent to use a T&E regimen after initial dosing.
* Treatment-naïve subjects for macular edema secondary to CRVO.
* Men and women ≥ 18 years of age.
* Documented BCVA of ETDRS letter score of 73 to 24 letters (Snellen equivalent of 20/40 to 20/320) in the study eye.

Exclusion Criteria:

* Previous PRP or macular laser photocoagulation in the study eye.
* Any prior or concomitant ocular treatment (e.g. anti-VEGF therapy, corticosteroids) in the study eye for macular edema secondary to RVO, except dietary supplements or vitamins prior to inclusion in the study. Intraocular anti-VEGF treatment is permitted for the treatment of diseases of fellow eye except for those that are specifically excluded.
* Prior systemic anti-VEGF or corticosteroid therapy, investigational or approved, within the last 3 months before the first dose in the study.
* Previous use of intraocular corticosteroids in the study eye at any time or use of periocular corticosteroids in the study eye within 12 months prior to Day 1.
* Any active intraocular, extraocular, and periocular inflammation or infection in either eye within 4 weeks of screening.
* Any history of allergy to povidone iodine.
* Known serious allergy to the fluorescein sodium for injection in angiography.
* Presence of any contraindications indicated in the EU commission/locally approved label for IVT aflibercept: hypersensitivity to the active substance IVT aflibercept or to any of the excipients; active or suspected ocular or periocular infection; active severe intraocular inflammation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2016-06-10 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (39):
- Australia (3):
  - Albury, New South Wales
  - Sydney, New South Wales
  - Parramatta
- Canada (6):
  - Calgary, Alberta
  - Hamilton, Ontario
  - London, Ontario
  - Boisbriand, Quebec
  - Sherbrooke, Quebec
  - Québec
- Denmark (2):
  - Aalborg
  - Glostrup Municipality
- France (3):
  - Bordeaux
  - Dijon
  - Lyon
- Germany (10):
  - Freiburg im Breisgau, Baden-Wurttemberg
  - Heidelberg, Baden-Wurttemberg
  - Karlsruhe, Baden-Wurttemberg
  - Augsburg, Bavaria
  - Göttingen, Lower Saxony
  - Cologne, North Rhine-Westphalia
  - Düsseldorf, North Rhine-Westphalia
  - Hannover, North Rhine-Westphalia
  - Münster, North Rhine-Westphalia
  - Leipzig, Saxony
- Italy (5):
  - Rome, Lazio
  - Milan, Lombardy
  - Ancona, The Marches
  - Pisa, Tuscany
  - Padua, Veneto
- Spain (4):
  - Sant Cugat Del Vallés, Barcelona
  - Viladecans, Barcelona
  - Oviedo, Principality of Asturias
  - Barcelona
- United Kingdom (6):
  - Sunderland, Tyne and Wear
  - Bradford, West Yorkshire
  - Bristol
  - Colchester
  - Liverpool
  - Oxford

REFERENCES:
- [Derived] Korobelnik JF, Larsen M, Eter N, Bailey C, Wolf S, Schmelter T, Allmeier H, Chaudhary V. Efficacy and Safety of Intravitreal Aflibercept Treat-and-Extend for Macular Edema in Central Retinal Vein Occlusion: the CENTERA Study. Am J Ophthalmol. 2021 Jul;227:106-115. doi: 10.1016/j.ajo.2021.01.027. Epub 2021 Feb 6. PMID 33556381
- See also: Click here to find results for studies related to Bayer products. — http://clinicaltrials.bayer.com/
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe — http://www.clinicaltrialsregister.eu/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 244 participants were screened in 42 study centers in 8 countries, the first subject first visit was on 10/Jun/2016 and last subject last visit was on 31/Jun/2019
Pre-assignment Details: Of the 244 screened participants, 162 subjects completed screening and entered the treatment period
Groups:
- Intravitreal (IVT) Aflibercept: Participants with macular edema secondary to CRVO were treated with 2 mg study drug intravitreal aflibercept over a treatment period of 76 weeks
Period: Overall Study
Arm/Group | Intravitreal (IVT) Aflibercept
Started | 162
Completed | 137
Not Completed | 25
Not completed — Death | 3
Not completed — Other | 10
Not completed — Physician Decision | 2
Not completed — Adverse Event | 6
Not completed — Withdrawal by Subject | 3
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Population: Safety analysis set: all participants who received any study drug
Arm/Group | Intravitreal (IVT) Aflibercept
Number analyzed (Participants) | 162
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.4 (13.3) [lower limit 13.3]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65
  Male | 97
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 156
  Unknown or Not Reported | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 154
  More than one race | 0
  Unknown or Not Reported | 4

OUTCOME MEASURES:

1. Secondary Outcome: The Mean Treatment Interval Between Injections
Time Frame: From baseline to Week 76
Population: Participants in full analysis set (received any study drug, had a baseline BCVA assessment and at least one post-baseline BCVA assessment) that completed study
Measure: Mean (Standard Deviation); unit: weeks
Arm/Group | Intravitreal (IVT) Aflibercept
Number analyzed (Participants) | 150
weeks | 6.37 (1.150) [lower limit 1.150]

2. Primary Outcome: The Proportion of Participants Who Gained ≥ 15 Letters in Best Corrected Visual Acuity (BCVA) on the Early Treatment Diabetic Retinopathy Score (ETDRS) Chart Compared to Baseline
Description: Participants who completed the study with a gain of ≥ 15 letters or dropped the study after Week 24 and having a permanent resolution of macular edema and a gain of ≥ 15 letters from baseline with regard to the latest BCVA assessment. The ETDRS chart includes 70 letters in total, more letters read correctly represents a better visual acuity.
Time Frame: Baseline, Week 24 and Week 76
Population: Full analysis set: included all participants who received any study drug, had a baseline BCVA assessment, and had at least one post-baseline BCVA assessment. Last observation carried forward (LOCF) imputation method.
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Intravitreal (IVT) Aflibercept
Number analyzed (Participants) | 160
percent | 65.6 (57.7) [57.7 to 72.9]
Statistical Analysis 1: Comparison: Intravitreal (IVT) Aflibercept; The null hypothesis "the proportion of participants with a ≥ 15-letter gain in BCVA at Week 76 is ≤ 40%" on the 2.5% level of significance (one-sided) was performed using the following criterion: If the p value is less than 2.5%, the null hypothesis will be rejected. Otherwise, the null hypothesis will be regarded as not rejected and may still be true; Test type: Other; p < 0.0001, Exact one-sided 1-sample binomial test

3. Primary Outcome: The Proportion of Participants With a Mean Treatment Interval Between Injections of ≥ 8 Weeks
Description: Participants who completed the study with a mean treatment interval between injections of ≥ 8 weeks or dropped out of the study after Week 24 and having a permanent resolution of macular edema
Time Frame: From the last actual visit of the initiation phase to Week 76
Population: Full analysis set: included all participants who received any study drug, had a baseline BCVA assessment, and had at least one post-baseline BCVA assessment
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Intravitreal (IVT) Aflibercept
Number analyzed (Participants) | 160
percent | 45.0 (37.1) [37.1 to 53.1]
Statistical Analysis 1: Comparison: Intravitreal (IVT) Aflibercept; The null hypothesis "the proportion of participants with a mean treatment interval of ≥ 8 weeks is ≤ 50%" on the 2.5% level of significance (one-sided) was performed using the following criterion: If the p value is less than 2.5%, the null hypothesis will be rejected. Otherwise, the null hypothesis will be regarded as not rejected and may still be true; Test type: Other; p = 0.8822, Exact one-sided 1-sample binomial test

4. Secondary Outcome: The Change in Best Corrected Visual Acuity (BCVA) as Measured by the Early Treatment Diabetic Retinopathy Letter Score (ETDRS) From Baseline
Description: The ETDRS chart includes 70 letters in total and the letter score ranges from 0 to 100. More letters read correctly results in a higher letter score, which represents better visual acuity
Time Frame: Baseline and Week 24, 52, and 76
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: scores
Arm/Group | Intravitreal (IVT) Aflibercept
Number analyzed (Participants) | 160
scores
  Absolute BCVA letter score at baseline | 51.9 (16.8) [lower limit 16.8]
  Absolute BCVA letter score at Week 24 | 72.4 (16.6) [lower limit 16.6]
  Absolute BCVA letter score at Week 52 | 71.8 (18.1) [lower limit 18.1]
  Absolute BCVA letter score at Week 76 | 72.3 (18.5) [lower limit 18.5]
  Change from baseline at Week 24 | 20.4 (17.0) [lower limit 17.0]
  Change from baseline at Week 52 | 19.9 (19.1) [lower limit 19.1]
  Change from baseline at Week 76 | 20.3 (19.5) [lower limit 19.5]

5. Secondary Outcome: The Change in Central Retinal Thickness (CRT) From Baseline
Description: CRT was measured in the study eye by spectral domain optical coherence tomography (SD-OCT).
Time Frame: Baseline and Week 24, 52 and 76
Population: Included all participants who received any study drug, had a baseline CRT assessment, and had post-baseline CRT assessment at Week 24, 52 and 76
Measure: Mean (Standard Deviation); unit: micrometer
Arm/Group | Intravitreal (IVT) Aflibercept
Number analyzed (Participants) | 158
micrometer
  Absolute CRT at baseline | 759.9 (246.0) [lower limit 246.0]
  Absolute CRT at Week 24 | 271.2 (53.1) [lower limit 53.1]
  Absolute CRT at Week 52 | 279.8 (106.8) [lower limit 106.8]
  Absolute CRT at Week 76 | 265.4 (57.9) [lower limit 57.9]
  Change from baseline at Week 24 | -488.9 (254.6) [lower limit 254.6]
  Change from baseline at Week 52 | -481.3 (266.5) [lower limit 266.5]
  Change from baseline at Week 76 | -496.1 (252.4) [lower limit 252.4]

6. Secondary Outcome: The Number of Injections Per Participant
Time Frame: From baseline to Week 76
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: injections
Arm/Group | Intravitreal (IVT) Aflibercept
Number analyzed (Participants) | 160
injections | 12.2 (2.53) [lower limit 2.53]

7. Secondary Outcome: The Proportion of Participants Who Gain ≥ 15 Letters in Best Corrected Visual Acuity (BCVA) on the Early Treatment Diabetic Retinopathy Score (ETDRS) Chart Compared to Baseline
Description: The ETDRS chart includes 70 letters in total. More letters read correctly represents a better visual acuity
Time Frame: Baseline and Week 24, Week 52
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Intravitreal (IVT) Aflibercept
Number analyzed (Participants) | 160
percent
  Week 24 | 68.8 (61.0) [61.0 to 75.8]
  Week 52 | 68.1 (60.3) [60.3 to 75.3]

8. Secondary Outcome: The Proportion of Participants With Change in Retinal Non-perfusion (FA/FP) Status From Baseline
Description: The change in retinal non-perfusion status by fundus angiography (FA)/fundus photography (FP)-confirmed ischemic disc area. The status was categorized into: no non-perfusion, <10 ischemic disc area, >=10 ischemic disc area and missing status
Time Frame: Baseline and Week 24, 52 and 76
Population: as for outcome 3
Measure: Number; unit: percent
Arm/Group | Intravitreal (IVT) Aflibercept
Number analyzed (Participants) | 160
percent
  Baseline to week 24: no to <10 | 4.4
  Baseline to week 24: no to >=10 | 3.8
  Baseline to week 24: no to missing | 6.3
  Baseline to week 24: <10 to no | 0.6
  Baseline to week 24: <10 to >=10 | 0.6
  Baseline to week 24: <10 to missing | 0
  Baseline to week 24: >=10 to no | 1.3
  Baseline to week 24: >=10 to <10 | 0
  Baseline to week 24: >=10 to missing | 0.6
  Baseline to week 24: missing to no | 0
  Baseline to week 24: missing to <10 | 0.6
  Baseline to week 24: missing to >=10 | 0.6
  Baseline to week 24: no status change | 81.9
  Baseline to week 52: no to <10 | 5.0
  Baseline to week 52: no to >=10 | 5.6
  Baseline to week 52: no to missing | 10.6
  Baseline to week 52: <10 to no | 1.9
  Baseline to week 52: <10 to >=10 | 0
  Baseline to week 52: <10 to missing | 0
  Baseline to week 52: >=10 to no | 1.9
  Baseline to week 52: >=10 to <10 | 0
  Baseline to week 52: >=10 to missing | 0
  Baseline to week 52: missing to no | 0
  Baseline to week 52: missing to <10 | 0.6
  Baseline to week 52: missing to >=10 | 0.6
  Baseline to week 52: no status change | 73.8
  Baseline to week 76: no to <10 | 3.1
  Baseline to week 76: no to >=10 | 4.4
  Baseline to week 76: no to missing | 18.1
  Baseline to week 76: <10 to no | 1.3
  Baseline to week 76: <10 to >=10 | 0.6
  Baseline to week 76: <10 to missing | 0.6
  Baseline to week 76: >=10 to no | 0.3
  Baseline to week 76: >=10 to <10 | 0
  Baseline to week 76: missing to no | 0
  Baseline to week 76: missing to <10 | 0.6
  Baseline to week 76: missing to >=10 | 0.6
  Baseline to week 76: no status change | 69.4

9. Secondary Outcome: The Proportion of Participants With Absence of Subretinal Fluid
Time Frame: Baseline, week 24, week 52 and week 76
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Intravitreal (IVT) Aflibercept
Number analyzed (Participants) | 160
percent
  Baseline | 25.6 [19.1 to 33.1]
  Week 24: number analyzed (Participants) | 154
  Week 24 | 98.7 [95.4 to 99.8]
  Week 52: number analyzed (Participants) | 153
  Week 52 | 95.4 [90.8 to 98.1]
  Week 76: number analyzed (Participants) | 137
  Week 76 | 97.8 [93.7 to 99.5]

10. Secondary Outcome: Incidence and Severity of Ocular Treatment-emergent Adverse Events
Time Frame: Up to 30 days after week 76
Population: Safety analysis set: included all participants who received any study drug
Measure: Count of Participants; unit: Participants
Arm/Group | Intravitreal (IVT) Aflibercept
Number analyzed (Participants) | 162
Participants
  Any ocular TEAEs | 90
  Severity: mild | 39
  Severity: moderate | 43
  Severity: severe | 8

ADVERSE EVENTS:
Time Frame: Up to 30 days after week 76
Arm/Group | Intravitreal (IVT) Aflibercept
All-Cause Mortality (participants affected / at risk) | 4/162
Serious Adverse Events (participants affected / at risk) | 32/162
Other Adverse Events (participants affected / at risk) | 81/162
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intravitreal (IVT) Aflibercept (N=162)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 4 (4)
Atrial flutter (Cardiac disorders) | 1 (1)
Bundle branch block bilateral (Cardiac disorders) | 1 (1)
Cardiac failure acute (Cardiac disorders) | 1 (1)
Mitral valve incompetence (Cardiac disorders) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 1 (1)
Amaurosis fugax (Eye disorders) | 1 (1)
Cataract (Eye disorders) | 1 (1)
Iridocyclitis (Eye disorders) | 1 (1)
Retinal artery occlusion (Eye disorders) | 1 (1)
Retinal degeneration (Eye disorders) | 1 (1)
Retinal ischaemia (Eye disorders) | 2 (2)
Retinal vein occlusion (Eye disorders) | 1 (1)
Visual acuity reduced (Eye disorders) | 1 (1)
Visual impairment (Eye disorders) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 2 (2)
Inguinal hernia (Gastrointestinal disorders) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1)
Hepatic haemorrhage (Hepatobiliary disorders) | 1 (1)
Endocarditis (Infections and infestations) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 1 (1)
Gastrointestinal viral infection (Infections and infestations) | 1 (1)
Urosepsis (Infections and infestations) | 1 (2)
Pneumonia (Infections and infestations) | 1 (1)
Latent syphilis (Infections and infestations) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Dementia (Nervous system disorders) | 1 (1)
Delirium (Psychiatric disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Renal colic (Renal and urinary disorders) | 1 (1)
Endometriosis (Reproductive system and breast disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1)
Haematoma (Vascular disorders) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intravitreal (IVT) Aflibercept (N=162)
Macular oedema (Eye disorders) | 12 (13)
Conjunctival haemorrhage (Eye disorders) | 18 (23)
Retinal ischaemia (Eye disorders) | 13 (16)
Retinal haemorrhage (Eye disorders) | 14 (14)
Visual acuity reduced (Eye disorders) | 26 (37)
Vitreous detachment (Eye disorders) | 9 (11)
Foreign body sensation in eyes (Eye disorders) | 9 (13)
Nasopharyngitis (Infections and infestations) | 26 (40)
Intraocular pressure increased (Investigations) | 20 (40)
Hypertension (Vascular disorders) | 19 (25)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2016-04-20): https://cdn.clinicaltrials.gov/large-docs/42/NCT02800642/Prot_000.pdf
  • Statistical Analysis Plan (2019-11-14): https://cdn.clinicaltrials.gov/large-docs/42/NCT02800642/SAP_001.pdf